CLINICAL TRIAL: NCT06849037
Title: and Infectious Morbidity Among Women With Meconium-stained Amniotic Fluid at Term, Between Those Who Will be Treated With Prophylactic Antibiotics Zinacef vs. Placebo
Brief Title: Comparing Infectious Morbidity Among Women With Meconium-stained Amniotic Fluid at Term, Between Those Treated With Prophylactic Antibiotics Zinacef vs. Placebo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Head of Maternal and Fetal medicine unit, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHR-0242-24; MOH_2025-01-30_013876 (Other: MOH-Israel)
Record Dates: First submitted 2025-02-15; First posted 2025-02-27 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Meconium-stained Amniotic Fluid; Chorioamnionitis
Keywords: meconium-stained amniotic fluid; antibiotic treatment; infectious morbidity; chorioamnionitis; zinacef
MeSH Terms: conditions — Chorioamnionitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinacef treatment (Experimental): women with meconium-stained amniotic fluid treated with zinacef 750 mg X3/d
  Interventions: Drug: zinacef tretment
- control (Placebo Comparator): women with meconium-stained amniotic fluid treated with I.V SALINE 100 CCX3/d
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: zinacef tretment — prophylactic antibiotic treatment with zinacef
  Arms: Zinacef treatment
Other: Placebo — I.V SALINE 100 CC X3/d
  Arms: control

SUMMARY:
Our randomized controlled double blind clinical trail aims to compare maternal and neonatal infectious morbidity between women with meconium-stained amniotic fluid treated with zinacef vs. placebo.

DETAILED DESCRIPTION:
The relationship between meconium staining and chorioamnionitis, as well as neonatal sepsis, has been documented, yet the precise mechanisms remain unclear. Additionally, the correlation between prolonged labor and meconium staining was described in the past. In light of these findings, our randomized controlled double blind trail aims to compare maternal and neonatal infectious morbidity between women with meconium-stained amniotic fluid treated with zinacef vs. placebo. Additionally, we aimed to assess the distribution of pathogens in chorioamnionitic swab cultures relative to the antibiotic treatment

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy at term
* meconium-stained amniotic fluid

Exclusion Criteria:

* Intrauterine fetal death
* GBS carriers
* zinacef allergy
* antibiotic treatment for other indication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnanct women
Enrollment: 182 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-02-13 (Estimated); Study Completion 2029-02-13 (Estimated)

PRIMARY OUTCOMES:
peripartum infections | 7 days
  chorioamnionitis and endometritis

SECONDARY OUTCOMES:
intrapartum fever | during labor up to 2 hours postpartum
  fever > 38
neonatal antibiotic treatment | 7 days
  antibiotic treatment
NICU admission | 1 week
  neonatal admission to the NICU after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Romero R, Hanaoka S, Mazor M, Athanassiadis AP, Callahan R, Hsu YC, Avila C, Nores J, Jimenez C. Meconium-stained amniotic fluid: a risk factor for microbial invasion of the amniotic cavity. Am J Obstet Gynecol. 1991 Mar;164(3):859-62. doi: 10.1016/0002-9378(91)90529-z. PMID 1900664
- [Background] Attali I, Korb D, Azria E, Lepercq J, Goffinet F, Schmitz T; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Meconium-stained amniotic fluid and neonatal morbidity in nulliparous patients with prolonged pregnancy. Acta Obstet Gynecol Scand. 2023 Aug;102(8):1092-1099. doi: 10.1111/aogs.14619. Epub 2023 Jun 28. PMID 37377254
- [Background] Rodriguez Fernandez V, Lopez Ramon Y Cajal CN, Marin Ortiz E, Couceiro Naveira E. Intrapartum and perinatal results associated with different degrees of staining of meconium stained amniotic fluid. Eur J Obstet Gynecol Reprod Biol. 2018 Sep;228:65-70. doi: 10.1016/j.ejogrb.2018.03.035. Epub 2018 Mar 20. PMID 29909265
- [Background] Addisu D, Asres A, Gedefaw G, Asmer S. Prevalence of meconium stained amniotic fluid and its associated factors among women who gave birth at term in Felege Hiwot comprehensive specialized referral hospital, North West Ethiopia: a facility based cross-sectional study. BMC Pregnancy Childbirth. 2018 Oct 30;18(1):429. doi: 10.1186/s12884-018-2056-y. PMID 30376814
- [Background] Gallo DM, Romero R, Bosco M, Gotsch F, Jaiman S, Jung E, Suksai M, Ramon Y Cajal CL, Yoon BH, Chaiworapongsa T. Meconium-stained amniotic fluid. Am J Obstet Gynecol. 2023 May;228(5S):S1158-S1178. doi: 10.1016/j.ajog.2022.11.1283. Epub 2023 Apr 1. PMID 37012128